CLINICAL TRIAL: NCT05176132
Title: South Danish Obesity Initiative (SDOI)
Brief Title: South Danish Obesity Initiative, Screening for Unrecognized Obesity Related Disease
Acronym: SDOI
Status: Recruiting | Type: Observational
Sponsor: Claus Bogh Juhl (Other)
Collaborators: Steno Diabetes Center Odense (Other); Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Claus Bogh Juhl, Professor, MD, PhD, Esbjerg Hospital - University Hospital of Southern Denmark
Organization: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Other Study IDs: SDOI
Record Dates: First submitted 2021-11-10; First posted 2022-01-04 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Obesity
Keywords: Obesity; Lifestyle intervention; BMI; Cohort; sleep apnea; diabetes; PCOS; NAFLD; Hypertension; Hyperlipidemia
MeSH Terms: conditions — Obesity; Sleep Apnea Syndromes; Diabetes Mellitus; Non-alcoholic Fatty Liver Disease; Hypertension; Hyperlipidemias | interventions — Self-Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood sample Feces sample Urine sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- OBESE (BMI>30): BMI above 30 kg/m2 and being 18 to 60 years of age. Since the initiative is open for the general obese population, the investigators did not define the size of the cohort, but expect around 500 referrals per year.
  Interventions: Other: Life style intervention (dietician+ physiotherapist); Other: Self management
- CONTROL Normal weight (BMI 20-25): 100 persons with normal weight (BMI 20 - 25 kg/m2) 18 to 60 years of age
  Interventions: Other: No intervention
- CONTROL Overweight (BMI 25-30): 100 persons with overweight (BMI 25 - 30 kg/m2) 18 to 60 years of age
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Life style intervention (dietician+ physiotherapist) — Obese patients with obesity related diseases will be invited to participate in a personalized lifestyle intervention program with dieticians and physiotherapists focusing on health improvement through personal motivation and perceived limitations and body accept.
  Groups: OBESE (BMI>30)
Other: Self management — Patients with no obesity related diseases will not be offered lifestyle intervention, but encouraged to physical activity (self management)
  Groups: OBESE (BMI>30)
Other: No intervention — Control groups (BMI 20-25 and BMI 25-30)
  Groups: CONTROL Normal weight (BMI 20-25); CONTROL Overweight (BMI 25-30)

SUMMARY:
People with BMI >30 kg/m2 will be included in at population-based cohort. Additionally, one control group with BMI 18.5-25 kg/m2 and one control group with BMI 25-30 kg/m2 will be included. All participants with age 18 and 60 years.

To evaluate health status participants will be screened by for undetected obesity-related diseases (hypertension, diabetes, dyslipidemia, sleep apnea, non-alcoholic fatty liver disease, chronic obstructive pulmonary disease, EKG-abnormalities, polycystic ovary syndrome (PCOS), and joint pain and for quality of life at baseline, 1 year, and 5 years. Additionally, anthropometric measurements are collected and a biobank is established for future research studies.

People with obesity related disease will be offered participation in a 12 month personalized lifestyle intervention program aimed at improvement of health and self-perception.

The collected data will be used to detect the prevalence for obesity-related disease to identify predictors for future obesity related disease and to evaluate the effect of a lifestyle intervention on health and quality of life.

DETAILED DESCRIPTION:
Obesity is associated with a variety of adverse health problems, and there is currently no effective scalable treatment with a durable effect. Additionally, well-known obesity related health problems are often underdiagnosed.

A Danish cohort of people with BMI >30 kg/m2 is established on University Hospital South West Jutland. Additionally, one control group with BMI 18.5-25 kg/m2 and one control group with BMI 25-30 kg/m2 will be included. Age range is defined as 18 and 60 years.

To evaluate health status all participants are screened by for undetected obesity-related diseases (hypertension, diabetes, dyslipidemia, sleep apnea, non-alcoholic fatty liver disease, chronic obstructive pulmonary disease, EKG-abnormalities, polycystic ovary syndrome (PCOS) and joint pain.

Data will be collected from questionnaires (Impact of Weight related on Quality of Life, Attitude to physical activity questionnaire, Adult Eating Behavior questionnaire, Berlin sleep apnea and Epworths Sleepiness scale, PCOS related questionnaire including Ferriman-Gallwey score, Work Ability Index, and weight history); clinical laboratory variables (HbA1c, glucose, c-peptide, lipid status, thyroid stimulating hormone (TSH), triiodothyronine (T3), thyroxine (T4), hemoglobin, thrombocytes, alanine aminotransferase (ALAT), aspartate aminotransferase (ASAT), bilirubin, gamma glutamic transferase, lactate dehydrogenase (LDH), alkaline phosphatase, and creatinine levels); and anthropometric measurements (blood pressure, EKG, liver elastography, spirometry (forced expiratory volume during first second as a fraction of forced vital capacity (FEV1/FVC), hand grip strength, gait speed, and CT scan for estimation of the subcutaneous and visceral fat volume). People with diseases uncovered by the screening program will be referred to specialized departments or general practice for further assessment and treatment.

A biobank (blood, feces, urine) is established for future research studies. Patients with obesity related diseases will be invited to participate in a personalized lifestyle intervention program with dietitians and physiotherapists focusing on health improvement through personal motivation, perceived limitations and body accept. Additionally, participants are invited to a 1 year follow-up. All participants, independent of disease status, will be invited for at new screening 5 years after the initial visit.

The data collected for the cohort will be used to estimate the prevalence and development of new obesity-related diseases, and to identify predictors for obesity-related diseases. Finally, the effect of the lifestyle intervention-program will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* BMI >30 (Obese cohort), BMI 20-25 (control group I), BMI 25-30 (control group II)
* Age 18-60 years

Exclusion Criteria:

* None

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants with BMI > 30 refered from 1) Genaral practice, 2) Other hospital Departments at Hosital South West Jutland, or 3) Psychiatric Department.
  The uptake area are 5 muncipalities with mixed urban and rural areas.
Sampling Method: Probability Sample
Enrollment: 2700 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of unrecognized obesity-related diseases | Baseline
  Undetected obesity-related diseases (hypertension, diabetes, dyslipidemia, sleep apnea, non-alcoholic fatty liver disease, chronic obstructive pulmonary disease, EKG-abnormalities, and polycystic ovary syndrome (PCOS).
Prevalence of unrecognized obesity-related diseases | 5 years
  Undetected obesity-related diseases (hypertension, diabetes, dyslipidemia, sleep apnea, non-alcoholic fatty liver disease, chronic obstructive pulmonary disease, EKG-abnormalities, and polycystic ovary syndrome (PCOS).

SECONDARY OUTCOMES:
Consultation systolic and diastolic blood pressure | Baseline
  Standard cut-of values
Consultation systolic and diastolic blood pressure | 1 year
  Standard cut-of values
Consultation systolic and diastolic blood pressure | 5 years
  Standard cut-of values
24 hour blood pressure | Baseline
  Measures mean blood pressure, day and night
24 hour blood pressure | 5 years
  Measures mean blood pressure, day and night
HbA1c | Baseline
  HbA1c equal to or higher than 48 mmol/mol indicates diabetes
HbA1c | 1 year
  HbA1c equal to or higher than 48 mmol/mol indicates diabetes
HbA1c | 5 years
  HbA1c equal to or higher than 48 mmol/mol indicates diabetes
Prediabetes | Baseline
  Hba1c 43-47 indicates prediabetes
Prediabetes | 1 year
  Hba1c 43-47 indicates prediabetes
Prediabetes | 5 years
  Hba1c 43-47 indicates prediabetes
Low density lipoprotein | Baseline
  Dyslipidemia is defined as low density lipoprotein (LDL) > 3 mmol/l or high density lipoprotein (HDL) cholesterol < 1 mmol/l.
Low density lipoprotein | 1 year
  Dyslipidemia is defined as low density lipoprotein (LDL) > 3 mmol/l or high density lipoprotein (HDL) cholesterol < 1 mmol/l.
Low density lipoprotein | 5 years
  Dyslipidemia is defined as low density lipoprotein (LDL) > 3 mmol/l or high density lipoprotein (HDL) cholesterol < 1 mmol/l.
Berlin sleep apnea questionnaire | Baseline
  Berlin sleep apnea questionnaire: The Berlin Questionnaire consists of three categories designed to elicit information regarding snoring (category 1), daytime somnolence (category 2), and the presence of obesity and/or hypertension (category 3). Categories 1 and 2 are considered positive if 2 or more responses are positive category 3 is considered positive if 1 response is positive and/or the body mass index is greater than 30 kg per meter squared. A patient is considered to have a high likelihood of sleep disordered breathing if 2 or more categories are positive.
Berlin sleep apnea questionnaire | 5 years
  Berlin sleep apnea questionnaire: The Berlin Questionnaire consists of three categories designed to elicit information regarding snoring (category 1), daytime somnolence (category 2), and the presence of obesity and/or hypertension (category 3). Categories 1 and 2 are considered positive if 2 or more responses are positive category 3 is considered positive if 1 response is positive and/or the body mass index is greater than 30 kg per meter squared. A patient is considered to have a high likelihood of sleep disordered breathing if 2 or more categories are positive.
Epworth Sleepiness Scale | Baseline
  Epworth Sleepiness Scale: Score 0-24. 0-5 Lower Normal Daytime Sleepiness, 6-10 Higher Normal Daytime Sleepiness, 11-12 Mild Excessive Daytime Sleepiness 13-15 Moderate Excessive Daytime Sleepiness, 16-24 Severe Excessive Daytime Sleepiness
Epworth Sleepiness Scale | 5 years
  Epworth Sleepiness Scale: Score 0-24. 0-5 Lower Normal Daytime Sleepiness, 6-10 Higher Normal Daytime Sleepiness, 11-12 Mild Excessive Daytime Sleepiness 13-15 Moderate Excessive Daytime Sleepiness, 16-24 Severe Excessive Daytime Sleepiness
Apnea hypopnoea index (AHI) | Baseline
  Quantifies sleep apnea cardiorespiratory monitoring: AHI < 5 per hour=normal or minimal, AHI ≥ 5, but < 15 per hour: mild, AHI ≥ 15, but < 30 per hour moderate and AHI ≥ 30 per hour: severe
Apnea hypopnoea index (AHI) | 5 years
  Quantifies sleep apnea cardiorespiratory monitoring: AHI < 5 per hour=normal or minimal, AHI ≥ 5, but < 15 per hour: mild, AHI ≥ 15, but < 30 per hour moderate and AHI ≥ 30 per hour: severe
Elastography | Baseline
  Quantifies liver-stiffness as a measure of non-alcoholic fatty liver disease, lower is better
Elastography | 5 years
  Quantifies liver-stiffness as a measure of non-alcoholic fatty liver disease, lower is better
FEV1/FVC | Baseline
  Indication of Chronic obstructive pulmonary disease as measured by spirometry
FEV1/FVC | 5 years
  Indication of Chronic obstructive pulmonary disease as measured by spirometry
EKG | Baseline
  Under resting conditions, standard 12 lead electrocardiography
EKG | 5 years
  Under resting conditions, standard 12 lead electrocardiography
Ferriman-Gallwey score self-reported | Baseline
  Measures hirsutism and indicates risk of Polycystic ovary syndrome (PCOS): Whole body equal or less than 10: normal, over 10: increased, Face: more than 2 is considered high and indicates hirsutism
Ferriman-Gallwey score self-reported | 5 years
  Measures hirsutism and indicates risk of Polycystic ovary syndrome (PCOS): Whole body equal or less than 10: normal, over 10: increased, Face: more than 2 is considered high and indicates hirsutism
Hand-grip force | Baseline
  Handgrip force: Higher is better, no defined cut-off value
Hand-grip force | 1 year
  Handgrip force: Higher is better, no defined cut-off value
Hand-grip force | five years
  Handgrip force: Higher is better, no defined cut-off value
Fat-free mass | Baseline
  Fat-free mass as estimated by bioimpedance measure, higher is better, no cut-of value
Fat-free mass | 1 year
  Fat-free mass as estimated by bioimpedance measure, higher is better, no cut-of value
Fat-free mass | 5 years
  Fat-free mass as estimated by bioimpedance measure, higher is better, no cut-of value
Gait-speed | Baseline
  Gait Speed in 6 meters: High more than 1.1 m/s, Median 0.7-1.1 m/s, Low <0.7 m/s
Gait-speed | 1 year
  Gait Speed in 6 meters: High more than 1.1 m/s, Median 0.7-1.1 m/s, Low <0.7 m/s
Gait-speed | 5 years
  Gait Speed in 6 meters: High more than 1.1 m/s, Median 0.7-1.1 m/s, Low <0.7 m/s
Body weight | Baseline
  Participants are weighed in light clothes with no shoes or pocket items, lower is better
Body weight | 1 year
  Participants are weighed in light clothes with no shoes or pocket items, lower is better
Body weight | 5 years
  Participants are weighed in light clothes with no shoes or pocket items, lower is better
BMI | Baseline
  Body weight / m2, lower is better
BMI | 1 year
  Body weight / m2, lower is better
BMI | 5 years
  Body weight / m2, lower is better
Waist circumference | Baseline
  Lower is better
Waist circumference | 1 year
  Lower is better
Waist circumference | 5 years
  Lower is better
Work-ability Index | Baseline
  Measures the ability of a person to work, higher values are better, no cut-of value
Work-ability Index | 5 years
  Measures the ability of a person to work, higher values are better, no cut-of value
Impact of weight on quality of life-lite | Baseline
  Measures weight associated quality of life, higher values are better, no cut-of value
Impact of weight on quality of life-lite | 1 year
  Measures weight associated quality of life, higher values are better, no cut-of value
Impact of weight on quality of life-lite | 5 years
  Measures weight associated quality of life, higher values are better, no cut-of value
Adult Eating Behavior Questionnaire | Baseline
  Measures eating behavior and appetite traits, descriptive
Adult Eating Behavior Questionnaire | 1 year
  Measures eating behavior and appetite traits, descriptive
Adult Eating Behavior Questionnaire | 5 years
  Measures eating behavior and appetite traits, descriptive
SDOI attitude to physical activity questionnaire | baseline
  Measures a persons attitude to physical activity, higher is better, no cut-of value
SDOI attitude to physical activity questionnaire | 1 year
  Measures a persons attitude to physical activity, higher is better, no cut-of value
SDOI attitude to physical activity questionnaire | 5 years
  Measures a persons attitude to physical activity, higher is better, no cut-of value

CONTACTS AND LOCATIONS:
Overall Officials: Claus B Juhl, Prof. PhD MD, Principal Investigator — Hospital South West Jutland, University hospital of Southern Denmark
Locations (1):
- Hospital of South West Jutland, University hospital of Southern Denmark, Esbjerg, Denmark

REFERENCES:
- [Derived] Juhl CB, Bladbjerg EM, Gram B, Knudsen T, Lauridsen MM, Nygaard NB, Drojdahl Ryg N, Skadhauge L, Munster AB. Prevalence of Obesity-Related Disease in a Danish Population - The Results of an Algorithm-Based Screening Program. Diabetes Metab Syndr Obes. 2024 Jun 19;17:2505-2517. doi: 10.2147/DMSO.S456028. eCollection 2024. PMID 38910914